CLINICAL TRIAL: NCT04241419
Title: A Pilot Study of High Intensity Walking in Older Adults in the Pre-operative Period
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unaware that the devices being used had a shelf life of only 6 months, the physical therapist could no longer assist with the study and did not have anyone to run the physical therapy aspect of the program.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB19-0468
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Frailty
Keywords: ESRD; Thoracic Disease; Kidney Transplant
MeSH Terms: conditions — Frailty; Kidney Failure, Chronic; Thoracic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Intensity Walking (Experimental): Participants will then undergo a 12 session intervention, with two sessions scheduled per week for six weeks. These will be 45 minute sessions, including 15 minutes of a warm-up and cool-down period as well as 30 minutes of walking. The intervention will include various types of over ground walking and stair work.
  Interventions: Behavioral: High Intensity Walking

INTERVENTIONS:
Behavioral: High Intensity Walking — Participants will then undergo a 12 session intervention, with two sessions scheduled per week for six weeks. These will be 45 minute sessions, including 15 minutes of a warm-up and cool-down period as well as 30 minutes of walking. The intervention will include various types of over ground walking and stair work.

SUMMARY:
The purpose of this pilot study is to evaluate a high intensity walking intervention in older surgical candidates with kidney or thoracic disease and pre-frailty or frailty.

DETAILED DESCRIPTION:
As the population ages, there are an increasing number of older adults presenting for surgical evaluation. Frailty evaluation has been recognized as a valuable tool in the pre-operative assessment of older adults. Frailty is a clinical syndrome with multiple causes and contributors that involves poor regulation of multiple physiologic systems and is characterized by reduced strength, endurance, and physiologic function. Frailty is a predictor of poor surgical outcomes in older patients, including post-operative complications, increased length of stay, post-discharge institutionalization, and mortality.Identification of frailty in the pre-operative period can aid in risk assessment and decision making for the procedure, can help inform a plan for post-operative care needs, and may provide a target for pre-operative risk reduction interventions.

Given the association of frailty with poor surgical outcomes and the high prevalence of frailty in surgical candidates, there has been much interest in interventions to mitigate this risk. Exercise interventions in other populations have shown success, although the optimal interventions are unknown. In both thoracic surgery and kidney transplantation, there may be a limited amount of time for intervention prior to the operation and patients often have other commitments, such as frequent medical appointments or dialysis sessions. Thus, a short duration program may be beneficial for these populations. High intensity walking is an approach that has shown to lead to functional gains in as short as 12 sessions. The therapists can also modify a high intensity walking program as needed for patients based on physical limitations, making it widely applicable for frail older adults of varying physical function levels, which is important to our older surgical populations. Surgical patients, which include kidney transplant and thoracic surgery patients, are particularly well suited to a pilot high intensity walking intervention given the high proportion of frailty and pre-frailty in these groups.

In this study, the investigator will examine a 12-week high intensity walking program for frail older surgical candidates.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Provision of informed consent
* No obvious contraindication to surgery such as uncontrolled cardiovascular, metabolic, or respiratory disease
* Have either thoracic disease that may require major surgery or End-Stage Renal Disease or Chronic Kidney Disease under consideration for kidney transplant. The kidney transplant patients enrolled must be either a candidate for living donor transplantation or on the expedited deceased donor kidney transplant list, which indicates they are expected to receive an offer in approximately the next 3-5 months.
* Able to ambulate at least 10 feet with moderate assistance (<50% physical assistance)
* Pre-frail or frail on the FRAIL screening tool (1+ positive on this tool)

Exclusion Criteria:

* Surgery planned within the 8 week study timeframe
* Uncontrolled cardiovascular, metabolic, or respiratory disease that limits exercise participation
* Resting blood pressure >180/110
* Any pre-existing health condition that would make the subject a poor candidate for this study in the opinion of the PI

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Phenotypic Frailty Criteria | 8 weeks
  The phenotypic frailty criteria is a validated frailty measurement tool. Phenotypic frailty is a composite that includes grip strength measured via a dynamometer, self-reported weight loss, self-reported exhaustion using a validated two question screen, 15 foot gait speed, and activity level measured by the Minnesota Leisure Time Physical Activity Questionnaire. This will be measured at baseline and 8 weeks.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | 8 weeks
  The SPPB is a mobility assessment which includes gait speed, sit to stand testing, and balance assessment. This will be measured at baseline and 8 weeks.
Berg Balance Scale | 8 weeks
  The Berg balance scale will be used to assess the subject's balance at baseline and 8 weeks.
6 minute walk test | 8 weeks
  The distance a subject can walk in 6 minutes will be measured at baseline and 8 weeks.
PROMIS Global Health | 8 weeks
  The PROMIS Global Health tool measures patient reported physical, mental, and social health, pain, and quality of life. This will be measured at baseline and 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Madariaga, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No